CLINICAL TRIAL: NCT01779726
Title: Efficiency of Diagnostic Strategy for Fast Track Lung Cancer Diagnosis. A Randomised Controlled Trial.
Brief Title: Efficiency of Diagnostic Strategy for Fast Track Lung Cancer Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 118/2011
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: Organization; of fast track
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT scan before chest physician (Experimental): CT scan before chest physician
  Interventions: Radiation: CT scan before chest physician
- Usual diagnostic workup (Active Comparator): Usual diagnostic workup
  Interventions: Radiation: Usual diagnostic workup

INTERVENTIONS:
Radiation: CT scan before chest physician — Patients referred to department of lung medicine are randomised according to the month of birth. Patients born in even months are CT scan before a consultation with a chest physician
  Arms: CT scan before chest physician
Radiation: Usual diagnostic workup — Patients born in odd months seen in the department of lung medicine by a chest physician and maybe then CT scanned (usual workup practice according to the fast track evaluation)
  Arms: Usual diagnostic workup

SUMMARY:
Annually, 4,200 new cases of lung cancer are diagnosed in Denmark. The stage of the disease is an important prognostic factor as an advanced stage reduces the opportunity for surgical intervention and other curative treatment. In denmark, as in many other countries, a fast track evaluation for lung cancer has been introduced in 2008.

When the general practitioners refer patients through the fast track, the majority of patients make their first visit to the Department of Pulmonary Medicine. After this visit, further investigation is initiated, which is often a CT scan of the chest and the upper abdomen. We dont know Whether this is the most appropriate organisation.

The aim of this project is to evaluate the way lung cancer patients are examined through the fast track and the impact of chest CT before an evaluation by a chest physician.

Investigators want to randomise all patients referred for the existing fast track to either direct CT scan of chest and upper abdomen or to evaluation by the chest physician, in order to test:

A) Fast track performance measured by number of CT scans and chest physician specialist time per diagnosis, and whether there is a difference between the intervention and the control group.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to fast track evaluation (lung department, Aarhus university hospital) from primary care.

Exclusion Criteria:

* Not referred from general practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Chest physician time | 2013
  Time (in minutes) spent by a chest physician pr patient

SECONDARY OUTCOMES:
Satisfaction with new organisation | 2013
  Measured with a qualitative focus interview with staff a the Department of lung medicine (doctors, nurses and secretary).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, M.D., Prof., Principal Investigator — The Research Unit for General Practice
Locations (2):
- Denmark (2):
  - Aarhus University, Aarhus, Aarhus
  - Department of lung medicine, Aarhus University Hospital, Aarhus, Aarhus

REFERENCES:
- [Derived] Guldbrandt LM, Fenger-Gron M, Folkersen BH, Rasmussen TR, Vedsted P. Reduced specialist time with direct computed tomography for suspected lung cancer in primary care. Dan Med J. 2013 Dec;60(12):A4738. PMID 24355447